CLINICAL TRIAL: NCT05128760
Title: Impact of Antiphospholipid Antibodies on Thrombin Generation During Sars-CoV2 Infection.
Brief Title: Impact of Antiphospholipid Antibodies on Thrombin Generation During Sars-CoV2 Infection (TACIT2 Study)
Acronym: TACIT2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Virginie Dufrost, Dr, Central Hospital, Nancy, France
Other Study IDs: 2021-A00244-37
Record Dates: First submitted 2021-11-18; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Antiphospholipid Syndrome; COVID-19
MeSH Terms: conditions — Antiphospholipid Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Patients with COVID-19 and aPL positivity: Patient with COVID-19 and aPL test positivity
  Interventions: Diagnostic Test: characterization of aPL
- Patients with COVID-19 without aPL positivity
  Interventions: Diagnostic Test: characterization of aPL
- APS patients
  Interventions: Diagnostic Test: characterization of aPL
- Healthy control
  Interventions: Diagnostic Test: characterization of aPL
- Disease control
  Interventions: Diagnostic Test: characterization of aPL

INTERVENTIONS:
Diagnostic Test: characterization of aPL — characterization of aPL profile, GT profile and leukocytes activations markers (NETs, TREM-1)

SUMMARY:
Context: Until 70% of thrombotic event are reported during Sars-CoV2 infection. Antiphospholipid antibodies (aPL) tests are often positive. We aim to determine if aPL positivity is involved in thrombose of Sars-CoV2 infection investigating the effect of aPL on thrombin generation (TG) and leucocyte pathway activation (neutrophils extracellular traps (NETs) and activation of triggering receptor expressed on myeloid cells 1 (TREM-1)).

Method: We will compare plasma from five groups of subjects: patients with antiphospholipid syndrome (APS) and patients hospitalized for Sars-CoV-2 infection with or without aPL, and as control, patients with acute venous thromboembolism event and healthy volunteers. For each subject, we will analyze aPL, activated protein C (APC) resistance measured by TG and leukocytes markers as circulating neutrophils extracellular traps (NETs) and soluble triggering receptor expressed on myeloid cells one (sTREM-1). We will control aPL test at three month and analyze their persistent positivity and association with thrombotic event.

Results: we hypothesize that patients with COVID-19 and aPL will have a similar aPL and level of APS resistance that patients with APS. Also, we think that circulating NETs and sTREM-1 levels will be more important in patients with COVID-19 with aPL than patients without aPL and similar in patients with COVID-19 and aPL and patients with APS.

Conclusion: our study will be the first to analyze the potential role of aPL on APC resistance measured by TG and neutrophil activation in COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving a comprehensive information about the study, and not opposed to participate

  + one criterion among :
* patient hospitalized fo a COVID-19
* Patient with known APS
* Patients hospitalized for an acute venous thromboembolism event aPL positivity or COVID-19
* healthy volunteers

Exclusion Criteria:

* For all participants : pregnancy, age below 18 years-old, absence of written informed consent , autoimmune or inflammatory disease except antiphospholipid syndrome
* For patients with COVID-19: previous aPL positivity (before COVID-19 infection)
* For patients with APS: previous symptomatic COVID-19 infection
* For patients control with acute venous thromboembolism event: previous symptomatic COVID-19 infection, infection or inflammatory disease in flare at the time of thromboembolism event, known aPL positivity
* For Healthy volunteers: history of thrombosis (venous, arterial or small vessels), previous symptomatic COVID-19 infection, infection or inflammatory disease in flare at the time of inclusion, known aPL positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Five groups of subjects will be enrolled in the study :
  1. patients hospitalized for à COVID-19 with aPL
  2. patients hospitalized for à COVID-19 without aPL
  3. patients with APS
  4. as control, patients with acute venous thromboembolism disease
  5. as control, healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of activated protein C resistance and comparison between groups | at inclusion

SECONDARY OUTCOMES:
frequency of positivity of each aPL test and comparison between groups | at inclusion
concentration of leucocytes activation markers and comparison between groups | at inclusion
frequency of persistent aPL test positivity and comparison between groups | at three month

CONTACTS AND LOCATIONS:
Overall Officials: Denis G Wahl, MD, PhD, Study Director — CHRU of Nancy; Stéphane Zuily, MD, PhD, Principal Investigator — CHRU of Nancy; Virginie Dufrost, MD, PhD, Principal Investigator — CHRU of Nancy
Locations (1):
- Virginie Dufrost, Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Bowles L, Platton S, Yartey N, Dave M, Lee K, Hart DP, MacDonald V, Green L, Sivapalaratnam S, Pasi KJ, MacCallum P. Lupus Anticoagulant and Abnormal Coagulation Tests in Patients with Covid-19. N Engl J Med. 2020 Jul 16;383(3):288-290. doi: 10.1056/NEJMc2013656. Epub 2020 May 5. No abstract available. PMID 32369280
- [Background] Zuily S, de Laat B, Guillemin F, Kelchtermans H, Magy-Bertrand N, Desmurs-Clavel H, Lambert M, Poindron V, de Maistre E, Dufrost V, Risse J, Shums Z, Norman GL, de Groot PG, Lacolley P, Lecompte T, Regnault V, Wahl D. Anti-Domain I beta2-Glycoprotein I Antibodies and Activated Protein C Resistance Predict Thrombosis in Antiphospholipid Syndrome: TAC(I)T Study. J Appl Lab Med. 2020 Nov 1;5(6):1242-1252. doi: 10.1093/jalm/jfaa072. PMID 32572467
- [Background] Yalavarthi S, Gould TJ, Rao AN, Mazza LF, Morris AE, Nunez-Alvarez C, Hernandez-Ramirez D, Bockenstedt PL, Liaw PC, Cabral AR, Knight JS. Release of neutrophil extracellular traps by neutrophils stimulated with antiphospholipid antibodies: a newly identified mechanism of thrombosis in the antiphospholipid syndrome. Arthritis Rheumatol. 2015 Nov;67(11):2990-3003. doi: 10.1002/art.39247. PMID 26097119
- [Background] Edel Y, Kliminski V, Pokroy-Shapira E, Oren S, Dortort Lazar A, Pri-Paz Basson Y, Egbaria M, Molad Y. Elevated plasma level of soluble triggering receptor expressed on myeloid cells-1 is associated with inflammation activity and is a potential biomarker of thrombosis in primary antiphospholipid syndrome. Arthritis Res Ther. 2019 Jan 7;21(1):10. doi: 10.1186/s13075-018-1779-5. PMID 30616644